CLINICAL TRIAL: NCT03235830
Title: Evaluation of Text Messaging as an Educational Method to Improve Healthcare Utilization
Brief Title: Text Messaging in Healthcare Utilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Matthew A. Broom, MD, FAAP, Associate Professor of Pediatrics, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 25160
Record Dates: First submitted 2017-07-30; First posted 2017-08-01 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Text Messaging
Keywords: Healthcare utilization; Health literacy

STUDY DESIGN:
Intervention Model Description: Caregivers of newborns (0-10 weeks of age) whose child received primary care at an urban, academic primary care clinic were approached for participation. Inclusion required reliable cellular and text messaging service and the ability to speak English. At intake, caregivers completed a brief demographic survey and were given a researcher-administered health literacy test called the Newest Vital Sign (NVS).
  Following the initial visit where consent, demographic information, and the NVS were obtained, participants were randomly assigned, by computer, to one of two groups: (1) caregiver receives only enhanced standard of care documents (ESoC), or (2) caregiver receives text messages in addition to enhanced standard of care documents (ESoC + Text). Both research team members and participants were blind to group assignment at the time of consent and enrollment. Clinic staff and providers were not aware of group assignment unless revealed by the participant.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Following the initial visit where consent, demographic information, and the NVS were obtained, participants were randomly assigned, by computer, to one of two groups: (1) caregiver receives only enhanced standard of care documents (ESoC), or (2) caregiver receives text messages in addition to enhanced standard of care documents (ESoC + Text). Both research team members and participants were blind to group assignment at the time of consent and enrollment. Clinic staff and providers were not aware of group assignment unless revealed by the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Standard of Care (ESoC) (Active Comparator): Subjects received a condensed version of the American Academy of Pediatrics Bright Futures content at their scheduled well-child visits though 6 months of age. The enhanced standard of care (ESoC) materials were added, by members of the research team, to registration packets and were given to caregivers by clinic staff, who were all trained to give the ESoC. For any patients who did not receive ESoC materials at their visit, an age-appropriate ESoC was mailed to the caregiver.
  Interventions: Behavioral: Enhanced Standard of Care (ESoC)
- Enhanced Standard of Care (ESoC) + Text (Experimental): Subjects assigned to the text messaging intervention group received four educational messages per week until their child was 6 months of age in addition to the ESoC documents. The text messages directly reflected Bright Futures and ESoC content, addressing infant development, safety, care, and the most common causes of nonurgent visits in the first year. Bright Futures content was adapted both for language and length to accommodate character limits and the patient population.
  Interventions: Behavioral: Enhanced Standard of Care (ESoC) + Text

INTERVENTIONS:
Behavioral: Enhanced Standard of Care (ESoC) + Text — See above in arm/group description
  Arms: Enhanced Standard of Care (ESoC) + Text
Behavioral: Enhanced Standard of Care (ESoC) — See above in arm/group description
  Arms: Enhanced Standard of Care (ESoC)

SUMMARY:
The overall goal is to assess the feasibility and effectiveness of using text messages as an educational tool in order to improve health care utilization among the parents and caregivers of newborns; in particular, the investigators seek to understand how educational text messages counteract the effects of low health literacy as it relates to non-urgent visits to the emergency department.

DETAILED DESCRIPTION:
Health care utilization is a issue germane to health care providers, insurers, and patients alike. Reducing non-urgent visits to the emergency department (ED) and primary care providers can improve both the quality and cost of care. There are barriers, however, to educating patients about more appropriate health care utilization. Low health literacy is one such barrier, particularly for caregivers of pediatric patients. Research reveals that up to half of caregivers seeking treatment at the ED have low levels of health literacy; levels that can make it more difficult to not only make sound decisions, but also provide effective follow-up care. Moreover, low levels of literacy perpetuate a cycle of seeking care for non-urgent conditions. Education initiatives designed to counteract the effects of low health literacy on health care utilization have been shown to reduce non-urgent ED visits by as much as 80%. These education interventions, while effective, are complex, costly, or time-intensive. For example, home visits by a nurse, parenting classes, and video tools are all shown to reduce non-urgent ED use, but each poses a unique problem for implementation in high volume, urban, pediatric primary care clinic. To date, no study has examined the effectiveness of text messaging as a possible avenue for educating caregivers about issues related to health care utilization. Text messaging has been shown to support behavioral change, and represents a fast and cost-effective alternative to more labor-intensive and expensive alternatives.

Danis Pediatrics, the pediatric practice of Saint Louis University physicians within SSM Cardinal Glennon Children's Medical Center (CGCMC), serves as a medical home to primarily urban, low-income patients. In the first half of 2014 alone, there were 5259 visits to the ED by caregivers of patients < 13 months of age. Of those, 520 Danis Pediatrics patients accounted for 919 of those visits. In short, just under 1 in 5 visits to the CGCMC ED is a Danis patient, and Danis patients visit the ED approximately 2 times in the first year. Previous studies of patients at Danis Pediatrics suggest that this population has access to text messaging and is interested in receiving healthcare-related information from their pediatric provider.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking parents and/or guardians of newborns (aged 0 to 2 months)
* Receive primary care at Danis Pediatrics
* Must have reliable mobile phone service and be able to receive text messages

Exclusion Criteria:

* Non-English speaking caregivers
* No reliable text messaging service

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2016-08-05 (Actual); Study Completion 2016-08-05 (Actual)

PRIMARY OUTCOMES:
Emergency department use | 6 months post end of intervention
  Number of emergency department visits

CONTACTS AND LOCATIONS:
Overall Officials: Matt Broom, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hodgkinson S, Godoy L, Beers LS, Lewin A. Improving Mental Health Access for Low-Income Children and Families in the Primary Care Setting. Pediatrics. 2017 Jan;139(1):e20151175. doi: 10.1542/peds.2015-1175. Epub 2016 Dec 12. PMID 27965378
- [Background] Yin HS, Johnson M, Mendelsohn AL, Abrams MA, Sanders LM, Dreyer BP. The health literacy of parents in the United States: a nationally representative study. Pediatrics. 2009 Nov;124 Suppl 3:S289-98. doi: 10.1542/peds.2009-1162E. PMID 19861483
- [Background] DeWalt DA, Hink A. Health literacy and child health outcomes: a systematic review of the literature. Pediatrics. 2009 Nov;124 Suppl 3:S265-74. doi: 10.1542/peds.2009-1162B. PMID 19861480
- [Background] Morrison AK, Schapira MM, Gorelick MH, Hoffmann RG, Brousseau DC. Low caregiver health literacy is associated with higher pediatric emergency department use and nonurgent visits. Acad Pediatr. 2014 May-Jun;14(3):309-14. doi: 10.1016/j.acap.2014.01.004. PMID 24767784
- [Background] DeAngelis C, Fosarelli P, Duggan AK. Use of the emergency department by children enrolled in a primary care clinic. Pediatr Emerg Care. 1985 Jun;1(2):61-5. PMID 3843434
- [Background] Salami O, Salvador J, Vega R. Reasons for nonurgent pediatric emergency department visits: perceptions of health care providers and caregivers. Pediatr Emerg Care. 2012 Jan;28(1):43-6. doi: 10.1097/PEC.0b013e31823f2412. PMID 22193700
- [Background] Morgan SR, Chang AM, Alqatari M, Pines JM. Non-emergency department interventions to reduce ED utilization: a systematic review. Acad Emerg Med. 2013 Oct;20(10):969-85. doi: 10.1111/acem.12219. PMID 24127700
- [Background] Yoffe SJ, Moore RW, Gibson JO, Dadfar NM, McKay RL, McClellan DA, Huang TY. A reduction in emergency department use by children from a parent educational intervention. Fam Med. 2011 Feb;43(2):106-11. PMID 21305425
- [Background] Fieldston ES, Nadel FM, Alpern ER, Fiks AG, Shea JA, Alessandrini EA. Effects of an education and training intervention on caregiver knowledge of nonurgent pediatric complaints and on child health services utilization. Pediatr Emerg Care. 2013 Mar;29(3):331-6. doi: 10.1097/PEC.0b013e31828512c7. PMID 23426249
- [Background] Zandieh SO, Gershel JC, Briggs WM, Mancuso CA, Kuder JM. Revisiting predictors of parental health care-seeking behaviors for nonurgent conditions at one inner-city hospital. Pediatr Emerg Care. 2009 Apr;25(4):238-243. doi: 10.1097/pec.0b013e31819e350e. PMID 19382324

DOCUMENTS (3):
  • Informed Consent Form (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT03235830/ICF_000.pdf
  • Study Protocol (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT03235830/Prot_001.pdf
  • Statistical Analysis Plan (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT03235830/SAP_002.pdf